CLINICAL TRIAL: NCT06248060
Title: Comparison and Opinion on the Safety of Teleconsultation
Brief Title: Comparison and Opinion on the Safety of Teleconsultation Versus Traditional Anaesthetic Consultation in a Day Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Céline Boudart, Principal Investigator, Erasme University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SRB2023303
Record Dates: First submitted 2024-01-26; First posted 2024-02-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pre-anaesthetic Consultation

STUDY DESIGN:
Intervention Model Description: Before - After study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before preanaesthetic teleconsultation implementation (Active Comparator)
  Interventions: Other: preanaesthetic classical physical consultation
- After preanaesthetic teleconsultation implementation (Experimental)
  Interventions: Other: preanaesthetic teleconsultation

INTERVENTIONS:
Other: preanaesthetic classical physical consultation — Pre-anaesthetic classical consultation before teleconsultation implementation
  Arms: Before preanaesthetic teleconsultation implementation
Other: preanaesthetic teleconsultation — Pre-anaesthetic consultation by telephone for eligible patients according to the criteria set
  Arms: After preanaesthetic teleconsultation implementation

SUMMARY:
A pre-anaesthetic consultation is compulsory. It must be carried out at least 8 days before a scheduled medical and/or surgical operation. Its main objectives are to take the patient's history, carry out a clinical examination, select the complementary examinations that should be carried out, and inform the patient of the procedure and the type of anaesthetic proposed. In a world moving towards virtualisation, a number of medical specialities have opted for remote consultations, either by telephone or video-conferencing. Teleconsultation seems to offer greater satisfaction, not only for patients, but also for surgeons and anaesthetists. It is also associated with a reduction in the distance travelled by patients, costs and financial expenditure, with no increase in the rate of cancellation of surgery. For the first time at the Brussels University Hospital (Erasme), the anaesthesia and intensive care team will gradually introduce the system of pre-anaesthetic teleconsultation by telephone from October 2023.

The aim of our study is to evaluate the effectiveness of preanaesthetic teleconsultation at the Erasme HUB. In fact, it would be better to have results based on local expertise in order to give an answer on the effectiveness, safety and security of this innovative method, which will be officially implemented in October 2023.

ELIGIBILITY:
Inclusion Criteria for prospective group (AFTER):

* Patients scheduled for any surgery at one day hospital and who have signed the consent form.
* Pre-anaesthetic consultation by telephone.

Inclusion Criteria for retrospective group (BEFORE):

* patients having undergone any surgery at one day hospital during the period between 01/01/2023 and 31/06/2023.
* Pre-anaesthetic consultation carried out face-to-face.
* Patients eligible for teleconsultation

Exclusion Criteria:

* Participation in another clinical study within the previous month.
* Patient unable to complete the questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Score of Patient endangerment (0-4) | at the 1 day of surgery
  Patient endangerment : 0 = Nothing to report; 1 = Lack of information but no danger to the patient; 2 =Lack of information and reduced safety but intervention maintained; 3 = Too great a risk to the patient.

SECONDARY OUTCOMES:
Satisfaction scores reported on LIKERT scale (1-5) | Baseline (before the procedure)
  How do you feel about the anaesthetic teleconsultation? 1 = Very satisfied; 2 = Satisfied; 3 = Neither satisfied nor dissatisfied; 4 = Not very satisfied; 5 = Not at all satisfied.
Pre-operative anxiety scorereported on LIKERT scale (1-5) | Baseline (before the procedure)
  How would you rate your level of anxiety? 1 = Not at all anxious; 2 = Slightly anxious; 3 = Moderately anxious; 4 = Somewhat anxious; 5 = Very anxious

CONTACTS AND LOCATIONS:
Overall Officials: boudart céline, Principal Investigator — HUB
Locations (1):
- Boudart Céline, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No